CLINICAL TRIAL: NCT05886647
Title: Non-invasive Neurostimulation and Rehabilitation in the Treatment of Patients With Respiratory Disorders: Randomized Controlled Clinical Trial
Brief Title: Non-invasive Neustimulation and Respiratory Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suellen Andrade (Other)
Responsible Party: Sponsor-Investigator, Suellen Andrade, Principal Investigator, Federal University of Paraíba
Organization: Federal University of Paraíba (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HD-tDCS+respiratory disorders
Record Dates: First submitted 2023-05-10; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Lung Diseases
Keywords: Brain Stimulation; Performance; Exercise
MeSH Terms: conditions — Lung Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 experimental (Experimental): group composed by patients with respiratory disorders, which will undergo 12 sessions of neurostimulation by HD-tDCS 4x1 (tDCS 1x1, developed by Soterix Medical Inc.).
  A current of 3 mA will be provided, positioning a central electrode (anode) on the left diaphragmatic primary motor cortex (4 cm lateral to the midline and 1 cm anterior to the binaural line) and the four return electrodes in a radius of 8 cm to the around. At the same time, inspiratory muscle training (IMT) will be performed by KH2; PowerBreathe International Ltd. UK with visual feedback, consisting of three series of two minutes of maximum and deep inspirations followed by two minutes of rest between them, totaling six minutes of TMI. The initial load will be through the maximum inspiratory pressure (MIP) achieved in the initial evaluation, using 40% of the total MIP in the first three weeks and 70% of the protocol will be used 40% of the MIP in the remaining three weeks and 70% in the remaining weeks.
  Interventions: Other: Active non-invasive stimulation and inspiratory muscle training
- Group 2 sham comparator (Sham Comparator): The participants allocated in the control group will receive the sham HD tDCS for 20 minutes associated with the IMT, following for this training the same load guidelines, duration and load increment used in the experimental group.
  Interventions: Other: Sham compatorator and inspiratory muscle training

INTERVENTIONS:
Other: Active non-invasive stimulation and inspiratory muscle training — Simultaneously with the current application, the patient will perform inspiratory muscle training (IMT) by KH2; PowerBreathe International Ltd. UK along with a feedback Breathelink, consisting of three series of two minutes of maximum and deep inspirations followed by two minutes of rest between them, totaling six minutes of TMI.
  Arms: Group 1 experimental
Other: Sham compatorator and inspiratory muscle training — As for the patients allocated in the control group, they will receive the HD-tDCS sham for 20 minutes associated with IMT, following for the same training, duration and load increment used in the experimental group.
  Arms: Group 2 sham comparator

SUMMARY:
Introduction: Respiratory diseases are associated with high rate of morbidity and mortality in Brazil. Cardiopulmonary rehabilitation through respiratory muscle training, aerobic training and strengthening of upper and lower limbs emerges as one of the resources available for the treatment and monitoring of patients with respiratory diseases. To add in this perspective, the application of HD-tDCS induces significant neurophysiological and clinical effects in several body systems.

Objective: To identify the chronic effects of non-invasive neurostimulation associated with the rehabilitation of patients with respiratory disorders. Material and methods: This is a pilot study, quantitative, clinical trial type, randomized and controlled, double blind. The sample will be composed by patients with respiratory diseases, aged above 18 years old. The study will consist of two groups: (1) HD-tDCS will be applied - anodic current + respiratory rehabilitation with respiratory muscle training (RMT) and (2) Sham - Only respiratory rehabilitation with RMT without any type of cortical stimulation. The chronic effects of neurostimulation by HD-tDCS associated with cardiopulmonary rehabilitation, with TMR, during 12 sessions will be evaluated. Patients will be evaluated, before and after the protocol, in relation to cortical activation function, pulmonary function, subjective perception of effort, respiratory muscle function, functional capacity, sensation of dyspnea and quality of life. For statistical analysis, intention-to-treat analysis will be used and groups will be compared using Student's t-test, for continuous variables, or chi-square, for categorical variables. ANOVA split-plot, repeated measures for primary outcomes. Analyzes of covariance to identify differences between groups using baseline scores as covariates. Effect sizes and confidence intervals will be calculated using eta squared (η²). Expected results: Neurostimulation would enhance the effects of respiratory rehabilitation and reduce the symptoms of patients with these diseases.

ELIGIBILITY:
Inclusion Criteria:

* confirmed clinical diagnosis for respiratory disease;
* stable disease

Exclusion Criteria:

* develop disabling condition that prevents the implementation of the protocol;
* join another rehabilitation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Lung function | six weeks
  Spirometry will be performed following the American Thoracic criteria Society (ATS). All participants will undergo a minimum of three maneuvers, in a sitting position, with a nose clip and mouthpiece attached. It will be instructed to perform maximum inspiration, up to total lung capacity, followed by a maximal and continuous forced expiration for at least six seconds, until residual volume.

SECONDARY OUTCOMES:
Maximum inspiratory pressure | six weeks
  To assess the maximum inspiratory pressure, a computerized electronic device (KH2; PowerBreathe International Ltd. United Kingdom) will be used. The participant will be seated, arms supported and nose clip to prevent air leaks.
  The maneuver consists of exhaling to the residual volume and performing a maximum inspiration maintained for as long as possible, being repeated 3 to 8 times to have a variation of less than 10%, based on the highest value.
functional capacity | six weeks
  Functional capacity will be assessed considering the distance covered in the six-minute walk test (6MWT). The 6MWT will be performed in a 30-meter corridor, checking heart rate (HR), peripheral oxygen saturation (SPO2), blood pressure (BP) and subjective perception of dyspnea by the Borg scale at the beginning and end of the test.
  HR and SpO2 will be observed throughout the test. For this porpuse, it will be used a stopwatch, a pulse oximeter to measure HR and SpO2, a sphygmomanometer to measure BP, a printed Borg scale that will be shown to the patient, a chair that can be moved to any area of the track and two cones to mark the return points that will be placed at the beginning and end of the test track.
  The test track will be marked in every 3 meters, in a closed environment and at a comfortable temperature.
  Instructions will be given for the patient to walk as fast as possible without running, in addition to warnings regarding the elapsed time of the test.
dyspnea sensation | six weeks
  For the evaluation of this outcome, it will be assessed by the dyspnea scale of the modified Medical Research Council (mMRC), which measures the degree of dyspnea in specific daily activities. The mMRC is divided into 4 grades, ranging from 0 (dyspnea on intense exercise) to 4 (dyspnea on minimal exertion) such as dressing or bathing). The scale is widely used in patients by its simplicity, easyness of use and correlation with quality of life, prognosis and distance covered in the six-minute walk test.
health-related quality of life | six weeks
  The assessment of health-related quality of life will be carried out through the application of a generic quality of life assessment questionnaire, the SF 36, which is a self-assessment instrument used to assess the quality of life of adults and is organized in eight dimensions: functionality (10 items), limitation caused by the physical problem (4 items), body pain (2 items), general health perception (5 items), vitality (4 items), social function (2 items), limitation caused by the emotional problem (3 items), mental health (5 items). A score is obtained through an algorithm (from 0 to 100), where 0 = lowest quality of life and 100 = better quality of life.
respiratory muscle resistance | six weeks
  To assess respiratory muscle resistance, a computerized electronic device (KH2; PowerBreathe International Ltd. United Kingdom) will be used. With the participant seated, arms supported and nose clip to prevent air leaks.
  The test consists of applying an incremental load, where the maximum number of breaths is performed for two minutes, starting with a load of 10 cmH2O and increasing this same value at each cycle, with a minute of rest. The highest value sustained for at least one minute will be considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Paraiba, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: will become available as it is collected, and will be available for a period of two years.

REFERENCES:
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Azabou E, Bao G, Heming N, Bounab R, Moine P, Chevallier S, Chevret S, Resche-Rigon M, Siami S, Sharshar T, Lofaso F, Annane D. Randomized Controlled Study Evaluating Efficiency of Low Intensity Transcranial Direct Current Stimulation (tDCS) for Dyspnea Relief in Mechanically Ventilated COVID-19 Patients in ICU: The tDCS-DYSP-COVID Protocol. Front Med (Lausanne). 2020 Jun 26;7:372. doi: 10.3389/fmed.2020.00372. eCollection 2020. PMID 32671084
- [Background] Bassi TG, Rohrs EC, Fernandez KC, Ornowska M, Nicholas M, Gani M, Evans D, Reynolds SC. Transvenous Diaphragm Neurostimulation Mitigates Ventilation-associated Brain Injury. Am J Respir Crit Care Med. 2021 Dec 15;204(12):1391-1402. doi: 10.1164/rccm.202101-0076OC. PMID 34491883
- [Background] Brunoni AR, Nitsche MA, Bolognini N, Bikson M, Wagner T, Merabet L, Edwards DJ, Valero-Cabre A, Rotenberg A, Pascual-Leone A, Ferrucci R, Priori A, Boggio PS, Fregni F. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. Brain Stimul. 2012 Jul;5(3):175-195. doi: 10.1016/j.brs.2011.03.002. Epub 2011 Apr 1. PMID 22037126
- [Background] Camargo LA, Pereira CA. Dyspnea in COPD: beyond the modified Medical Research Council scale. J Bras Pneumol. 2010 Sep-Oct;36(5):571-8. doi: 10.1590/s1806-37132010000500008. English, Portuguese. PMID 21085822
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Dias FD, Sampaio LM, da Silva GA, Gomes EL, do Nascimento ES, Alves VL, Stirbulov R, Costa D. Home-based pulmonary rehabilitation in patients with chronic obstructive pulmonary disease: a randomized clinical trial. Int J Chron Obstruct Pulmon Dis. 2013;8:537-44. doi: 10.2147/COPD.S50213. Epub 2013 Nov 5. PMID 24235824
- [Background] Dmochowski JP, Datta A, Bikson M, Su Y, Parra LC. Optimized multi-electrode stimulation increases focality and intensity at target. J Neural Eng. 2011 Aug;8(4):046011. doi: 10.1088/1741-2560/8/4/046011. Epub 2011 Jun 10. PMID 21659696
- [Background] Edwards D, Cortes M, Datta A, Minhas P, Wassermann EM, Bikson M. Physiological and modeling evidence for focal transcranial electrical brain stimulation in humans: a basis for high-definition tDCS. Neuroimage. 2013 Jul 1;74:266-75. doi: 10.1016/j.neuroimage.2013.01.042. Epub 2013 Jan 28. PMID 23370061
- [Background] Filipas L, Gallo G, Meloni A, Luzi L, Codella R. Effects of bilateral dorsolateral prefrontal cortex high-definition transcranial direct-current stimulation on time-trial performance in cyclists with type 1 diabetes mellitus. Brain Stimul. 2022 Sep-Oct;15(5):1292-1299. doi: 10.1016/j.brs.2022.09.005. Epub 2022 Sep 17. PMID 36126864
- [Background] Laviolette L, Nierat MC, Hudson AL, Raux M, Allard E, Similowski T. The supplementary motor area exerts a tonic excitatory influence on corticospinal projections to phrenic motoneurons in awake humans. PLoS One. 2013 Apr 16;8(4):e62258. doi: 10.1371/journal.pone.0062258. Print 2013. PMID 23614046
- [Background] Morya E, Monte-Silva K, Bikson M, Esmaeilpour Z, Biazoli CE Jr, Fonseca A, Bocci T, Farzan F, Chatterjee R, Hausdorff JM, da Silva Machado DG, Brunoni AR, Mezger E, Moscaleski LA, Pegado R, Sato JR, Caetano MS, Sa KN, Tanaka C, Li LM, Baptista AF, Okano AH. Beyond the target area: an integrative view of tDCS-induced motor cortex modulation in patients and athletes. J Neuroeng Rehabil. 2019 Nov 15;16(1):141. doi: 10.1186/s12984-019-0581-1. PMID 31730494
- [Background] Nakayama T, Fujii Y, Suzuki K, Kanazawa I, Nakada T. The primary motor area for voluntary diaphragmatic motion identified by high field fMRI. J Neurol. 2004 Jun;251(6):730-5. doi: 10.1007/s00415-004-0413-4. PMID 15311350
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Pereira CA, Sato T, Rodrigues SC. New reference values for forced spirometry in white adults in Brazil. J Bras Pneumol. 2007 Jul-Aug;33(4):397-406. doi: 10.1590/s1806-37132007000400008. English, Portuguese. PMID 17982531
- [Background] Pilloni G, Bikson M, Badran BW, George MS, Kautz SA, Okano AH, Baptista AF, Charvet LE. Update on the Use of Transcranial Electrical Brain Stimulation to Manage Acute and Chronic COVID-19 Symptoms. Front Hum Neurosci. 2020 Nov 12;14:595567. doi: 10.3389/fnhum.2020.595567. eCollection 2020. PMID 33281589
- [Background] Polkey MI, Moxham J. Attacking the disease spiral in chronic obstructive pulmonary disease. Clin Med (Lond). 2006 Mar-Apr;6(2):190-6. doi: 10.7861/clinmedicine.6-2-190. PMID 16688981
- [Background] Singer J, Yelin EH, Katz PP, Sanchez G, Iribarren C, Eisner MD, Blanc PD. Respiratory and skeletal muscle strength in chronic obstructive pulmonary disease: impact on exercise capacity and lower extremity function. J Cardiopulm Rehabil Prev. 2011 Mar-Apr;31(2):111-9. doi: 10.1097/HCR.0b013e3182033663. PMID 21240003
- [Background] Shields GS, Coissi GS, Jimenez-Royo P, Gambarota G, Dimber R, Hopkinson NS, Matthews PM, Brown AP, Polkey MI. Bioenergetics and intermuscular fat in chronic obstructive pulmonary disease-associated quadriceps weakness. Muscle Nerve. 2015 Feb;51(2):214-21. doi: 10.1002/mus.24289. Epub 2014 Nov 19. PMID 24831173
- [Background] Silva CMDSE, Gomes Neto M, Saquetto MB, Conceicao CSD, Souza-Machado A. Effects of upper limb resistance exercise on aerobic capacity, muscle strength, and quality of life in COPD patients: a randomized controlled trial. Clin Rehabil. 2018 Dec;32(12):1636-1644. doi: 10.1177/0269215518787338. Epub 2018 Jul 16. PMID 30012033
- [Background] Souza DUF, Monteiro DP, Pinto RZ, Pereira DAG. Supervised Exercise Therapy for Intermittent Claudication. Phys Ther. 2020 Jan 23;100(1):8-13. doi: 10.1093/ptj/pzz140. PMID 31612216
- [Background] Schulz KF, Altman DG, Moher D. CONSORT 2010 statement: Updated guidelines for reporting parallel group randomised trials. J Pharmacol Pharmacother. 2010 Jul;1(2):100-7. doi: 10.4103/0976-500X.72352. No abstract available. PMID 21350618
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Maltais F, Decramer M, Casaburi R, Barreiro E, Burelle Y, Debigare R, Dekhuijzen PN, Franssen F, Gayan-Ramirez G, Gea J, Gosker HR, Gosselink R, Hayot M, Hussain SN, Janssens W, Polkey MI, Roca J, Saey D, Schols AM, Spruit MA, Steiner M, Taivassalo T, Troosters T, Vogiatzis I, Wagner PD; ATS/ERS Ad Hoc Committee on Limb Muscle Dysfunction in COPD. An official American Thoracic Society/European Respiratory Society statement: update on limb muscle dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 May 1;189(9):e15-62. doi: 10.1164/rccm.201402-0373ST. PMID 24787074
- [Background] Foster C, Florhaug JA, Franklin J, Gottschall L, Hrovatin LA, Parker S, Doleshal P, Dodge C. A new approach to monitoring exercise training. J Strength Cond Res. 2001 Feb;15(1):109-15. PMID 11708692
- [Background] Barreiro E, Gea J. Respiratory and Limb Muscle Dysfunction in COPD. COPD. 2015 Aug;12(4):413-26. doi: 10.3109/15412555.2014.974737. PMID 25438125
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058